CLINICAL TRIAL: NCT06342115
Title: Ceftolozane/Tazobactam Versus Meropenem for Febrile Neutropenia on Patients Colonized With or at Risk for Infection With Extended Spectrum Beta Lactamase (ESBL)-Producing Pathogens: a Randomized Double-blind Non-inferiority Trial.
Brief Title: Ceftolozane/Tazobactam Versus Meropenem for Febrile Neutropenia on Patients Colonized With or at Risk for Infection With Extended Spectrum Beta Lactamase - Producing Pathogens
Acronym: CLEMENT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, João Antonio Gonçalves Garreta Prats, Principal Investigator, Beneficência Portuguesa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEMENT TRIAL
Record Dates: First submitted 2024-02-29; First posted 2024-04-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Febrile Neutropenia
Keywords: Febrile Neutropenia; Ceftolozane/tazobactam; ESBL; Meropenem
MeSH Terms: conditions — Febrile Neutropenia | interventions — ceftolozane, tazobactam drug combination; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the intervention arm 3g of ceftolozane-tazobactam are given intravenously every 8 hours. Duration of therapy should follow local guidelines and de-escalation is allowed after identification of causative pathogens.
  Colonized patients will be considered those identified through positive routine rectal swabs and/or positive culture of a clinical sample) or at risk of infection by an ESBL-producing pathogen due to use of 3rd/4th gen cephalosporin or piperacillin/tazobactam for at least 48 hours. in the last 30 days.
  Interventions: Drug: Ceftolozane-Tazobactam
- Control (Active Comparator): The comparator arm consists of 2g of meropenem given intravenously every 8 hours.Duration of therapy should follow local guidelines and de-escalation is allowed after identification of causative pathogens.
  Colonized patients will be considered those identified through positive routine rectal swabs and/or positive culture of a clinical sample) or at risk of infection by an ESBL-producing pathogen due to use of 3rd/4th gen cephalosporin or piperacillin/tazobactam for at least 48 hours. in the last 30 days.
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Ceftolozane-Tazobactam — In the intervention arm 3g of ceftolozane-tazobactam are given intravenously every 8 hours. Duration of therapy should follow local guidelines and de-escalation is allowed after identification of causative pathogens.
  Arms: Intervention
Drug: Meropenem — The comparator arm consists of 2g of meropenem given intravenously every 8 hours.Duration of therapy should follow local guidelines and de-escalation is allowed after identification of causative pathogens.
  Arms: Control

SUMMARY:
The study proposes a planned, double-blind, non-inferiority clinical trial involving patients with febrile neutropenia and risk of extended-spectrum beta-lactamase (ESBL) infection. The goal is:

- Analyze the efficacy and tolerability of Ceftolozane/tazobactam (CEF/TAZ) compared to the current standard of care (meropenem) in patients with febrile neutropenia and risk of ESBL infection.

Patients will be randomly assigned to receive CEF/TAZ or meropenem, with assessment of clinical response, toxicity and microbiological evolution. Stool samples will be collected before, during and after treatment for intestinal microbiota analysis and intestinal microbiome analysis to evaluate possible effects on GVHD. Analysis of the results will include the taxonomic classification of the organisms present. Data will be analyzed to assess non-inferiority in clinical response, incidence of GVHD, antimicrobial resistance and other outcomes.

ELIGIBILITY:
Inclusion criteria:

- Individuals who present with the onset of febrile neutropenia and at the same time present colonization with an ESBL-producing pathogen (identified through positive routine rectal swabs and/or positive culture of clinical specimen) or risk of infection with an ESBL-producing pathogen (use of 3rd/4th gen cephalosporin or piperacillin/tazobactam for at least 48 hours in the last 30 days).

Exclusion Criteria:

* Patients known to be colonized with carbapenem-resistant or CEF/TAZ-resistant pathogens
* Patients with previous use of carbapenems for at least 48h in the past 30 days are also excluded due to risk of resistance to the study drugs.
* Growth of a pathogen resistant to either study drug in a relevant clinical specimen during the intervention phase will be followed by adjustment of therapy according to local protocol, unblinding, and exclusion from the study.
* Patients that have received less than 72h of either study drug will also be excluded from the final analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 176 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Clinical Response of Clinical Cure at the End-of-Therapy (EOT) Visit in the Intent-to-Treat (ITT) Population | Within 24 hours after last dose of study drug (Up to ~Day 15)
  To compare the clinical response rates at the EOT visit for ceftolozane/tazobactam versus meropenem. Clinical response at the EOT visit was defined as cure (complete resolution of fever and symptoms related to Febrile Neutropenia episode), failure (non-resolution, relapse or recurrence of Febrile Neutropenia) or indeterminate (no evaluable study data). A favorable clinical response is a clinical cure. A missing clinical response will be considered indeterminate.

SECONDARY OUTCOMES:
Percentage of Participants With Clinical Response of Clinical Cure at the End-of-Therapy (EOT) Visit in the Microbiological Intent-to-Treat (mITT) Population | 7 to 14 days after last dose of study drug (Up to ~Day 30)
  To compare the clinical response rates at the EOT visit for ceftolozane/tazobactam versus meropenem in the Microbiological Intent-to-Treat (mITT) Population. Clinical response at the EOT visit was defined as cure (complete resolution of fever and symptoms related to Febrile Neutropenia episode), failure (non-resolution, relapse or recurrence of Febrile Neutropenia) or indeterminate (no evaluable study data). A favorable clinical response is a clinical cure. A missing clinical response will be considered indeterminate.
Percentage of Participants With Clinical Response of Clinical Cure at the Test-of-Cure (TOC) Visit in the Intent-to-Treat (ITT) Population | 7 to 14 days after last dose of study drug (Up to ~Day 30)
  To demonstrate the non-inferiority of ceftolozane/tazobactam versus meropenem in participants with Febrile Neutropenia on Patients Colonized With or at Risk for Infection With Extended Spectrum Beta Lactamase - Producing Pathogens at the TOC visit (7 to 14 days after the end-of-therapy [EOT] visit) using a non-inferiority margin of 12.5%. Clinical response at the TOC visit was defined as cure (complete resolution of fever and symptoms related to Febrile Neutropenia), failure (non-resolution, relapse or recurrence of Febrile Neutropenia) or indeterminate (no evaluable study data). A favorable clinical response is a clinical cure. A missing clinical response will be considered indeterminate unless the clinical outcome at the EOT visit was failure.
Incidence of microbiologically documented infections and identification of causative organisms in culture | Up to 100 days
  The incidences of microbiologically documented infections, along with the identification of causative organisms in culture, will be recorded. The measure will be assessed through the counting of cases confirmed by positive cultures.
In-hospital mortality | Until100 days after allogenic HSCT
  In-hospital mortality in the first 100 days after allogenic hematopoietic stem cell transplant (HSCT)
Occurrence of graft versus host disease (GVHD) | Until100 days after allogenic HSCT
  Occurrence of GVHD In the first 100 days after allogenic HSCT
Frequency of multidrug resistant-pathogen infections or colonization | Until100 days after allogenic HSCT
  Frequency of multidrug resistant-pathogen infections or colonization by weekly rectal swab screening
Faecal microbiota analysis | Up to 100 days
  Patients will also undergo faecal microbiota analysis on baseline and at the end of therapy as a surrogate marker for future GVHD.
Percentage of Participants Who Report 1 or More Adverse Event (AE) | Up to 35 days after last dose of study drug
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Percentage of Participants With Any Serious Adverse Event (SAE) | Up to 35 days after last dose of study drug (Up to ~Day 50) ]
  A serious adverse event (SAE) is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Percentage of Participants Discontinuing Study Drug Due to an Adverse Event (AE) | Up to 14 days after the first dose of study drug (Up to ~Day 15)
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: João Prats, MD, Principal Investigator — A Beneficência Portuguesa de São Paulo
Locations (1):
- A Beneficência Portuguesa de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pillinger KE, Bouchard J, Withers ST, Mediwala K, McGee EU, Gibson GM, Bland CM, Bookstaver PB. Inpatient Antibiotic Stewardship Interventions in the Adult Oncology and Hematopoietic Stem Cell Transplant Population: A Review of the Literature. Ann Pharmacother. 2020 Jun;54(6):594-610. doi: 10.1177/1060028019890886. Epub 2019 Nov 26. PMID 31771337
- [Background] Coates ARM, Hu Y, Holt J, Yeh P. Antibiotic combination therapy against resistant bacterial infections: synergy, rejuvenation and resistance reduction. Expert Rev Anti Infect Ther. 2020 Jan;18(1):5-15. doi: 10.1080/14787210.2020.1705155. PMID 31847614
- [Background] Meletis G. Carbapenem resistance: overview of the problem and future perspectives. Ther Adv Infect Dis. 2016 Feb;3(1):15-21. doi: 10.1177/2049936115621709. PMID 26862399
- [Background] Girmenia C, Rossolini GM, Piciocchi A, Bertaina A, Pisapia G, Pastore D, Sica S, Severino A, Cudillo L, Ciceri F, Scime R, Lombardini L, Viscoli C, Rambaldi A; Gruppo Italiano Trapianto Midollo Osseo (GITMO); Gruppo Italiano Trapianto Midollo Osseo GITMO. Infections by carbapenem-resistant Klebsiella pneumoniae in SCT recipients: a nationwide retrospective survey from Italy. Bone Marrow Transplant. 2015 Feb;50(2):282-8. doi: 10.1038/bmt.2014.231. Epub 2014 Oct 13. PMID 25310302
- [Background] Cattaneo C, Di Blasi R, Skert C, Candoni A, Martino B, Di Renzo N, Delia M, Ballanti S, Marchesi F, Mancini V, Orciuolo E, Cesaro S, Prezioso L, Fanci R, Nadali G, Chierichini A, Facchini L, Picardi M, Malagola M, Orlando V, Trecarichi EM, Tumbarello M, Aversa F, Rossi G, Pagano L; SEIFEM Group. Bloodstream infections in haematological cancer patients colonized by multidrug-resistant bacteria. Ann Hematol. 2018 Sep;97(9):1717-1726. doi: 10.1007/s00277-018-3341-6. Epub 2018 Apr 28. PMID 29705860
- [Background] Camargo JF, Anderson AD, Natori Y, Natori A, Morris MI, Pereira D, Komanduri KV. Early antibiotic use is associated with CMV risk and outcomes following allogeneic hematopoietic cell transplantation. Blood Adv. 2020 Dec 22;4(24):6364-6367. doi: 10.1182/bloodadvances.2020003277. No abstract available. PMID 33351132
- [Background] Tanaka JS, Young RR, Heston SM, Jenkins K, Spees LP, Sung AD, Corbet K, Thompson JC, Bohannon L, Martin PL, Stokhuyzen A, Vinesett R, Ward DV, Bhattarai SK, Bucci V, Arshad M, Seed PC, Kelly MS. Anaerobic Antibiotics and the Risk of Graft-versus-Host Disease after Allogeneic Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2020 Nov;26(11):2053-2060. doi: 10.1016/j.bbmt.2020.07.011. Epub 2020 Jul 17. PMID 32682948
- [Background] van Duin D, Bonomo RA. Ceftazidime/Avibactam and Ceftolozane/Tazobactam: Second-generation beta-Lactam/beta-Lactamase Inhibitor Combinations. Clin Infect Dis. 2016 Jul 15;63(2):234-41. doi: 10.1093/cid/ciw243. Epub 2016 Apr 20. PMID 27098166
- [Background] Gomis-Font MA, Cabot G, Lopez-Arguello S, Zamorano L, Juan C, Moya B, Oliver A. Comparative analysis of in vitro dynamics and mechanisms of ceftolozane/tazobactam and imipenem/relebactam resistance development in Pseudomonas aeruginosa XDR high-risk clones. J Antimicrob Chemother. 2022 Mar 31;77(4):957-968. doi: 10.1093/jac/dkab496. PMID 35084040
- [Background] Bitar I, Salloum T, Merhi G, Hrabak J, Araj GF, Tokajian S. Genomic Characterization of Mutli-Drug Resistant Pseudomonas aeruginosa Clinical Isolates: Evaluation and Determination of Ceftolozane/Tazobactam Activity and Resistance Mechanisms. Front Cell Infect Microbiol. 2022 Jun 15;12:922976. doi: 10.3389/fcimb.2022.922976. eCollection 2022. PMID 35782142
- [Background] Timsit JF, Huntington JA, Wunderink RG, Shime N, Kollef MH, Kivistik U, Novacek M, Rea-Neto A, Martin-Loeches I, Yu B, Jensen EH, Butterton JR, Wolf DJ, Rhee EG, Bruno CJ. Ceftolozane/tazobactam versus meropenem in patients with ventilated hospital-acquired bacterial pneumonia: subset analysis of the ASPECT-NP randomized, controlled phase 3 trial. Crit Care. 2021 Aug 11;25(1):290. doi: 10.1186/s13054-021-03694-3. PMID 34380538
- [Background] Solomkin J, Hershberger E, Miller B, Popejoy M, Friedland I, Steenbergen J, Yoon M, Collins S, Yuan G, Barie PS, Eckmann C. Ceftolozane/Tazobactam Plus Metronidazole for Complicated Intra-abdominal Infections in an Era of Multidrug Resistance: Results From a Randomized, Double-Blind, Phase 3 Trial (ASPECT-cIAI). Clin Infect Dis. 2015 May 15;60(10):1462-71. doi: 10.1093/cid/civ097. Epub 2015 Feb 10. PMID 25670823
- [Background] Wagenlehner FM, Umeh O, Steenbergen J, Yuan G, Darouiche RO. Ceftolozane-tazobactam compared with levofloxacin in the treatment of complicated urinary-tract infections, including pyelonephritis: a randomised, double-blind, phase 3 trial (ASPECT-cUTI). Lancet. 2015 May 16;385(9981):1949-56. doi: 10.1016/S0140-6736(14)62220-0. Epub 2015 Apr 27. PMID 25931244
- [Background] Chaftari AM, Hachem R, Malek AE, Mulanovich VE, Szvalb AD, Jiang Y, Yuan Y, Ali S, Deeba R, Chaftari P, Raad I. A Prospective Randomized Study Comparing Ceftolozane/Tazobactam to Standard of Care in the Management of Neutropenia and Fever in Patients With Hematological Malignancies. Open Forum Infect Dis. 2022 Feb 14;9(6):ofac079. doi: 10.1093/ofid/ofac079. eCollection 2022 Jun. PMID 35663286
- [Background] Clerici D, Oltolini C, Greco R, Ripa M, Giglio F, Mastaglio S, Lorentino F, Pavesi F, Farina F, Liberatore C, Castiglion B, Tassan Din C, Bernardi M, Corti C, Peccatori J, Scarpellini P, Ciceri F, Castagna A. The place of ceftazidime/avibactam and ceftolozane/tazobactam for therapy of haematological patients with febrile neutropenia. Int J Antimicrob Agents. 2021 Jun;57(6):106335. doi: 10.1016/j.ijantimicag.2021.106335. Epub 2021 Apr 7. PMID 33838223
- [Background] Bergas A, Albasanz-Puig A, Fernandez-Cruz A, Machado M, Novo A, van Duin D, Garcia-Vidal C, Hakki M, Ruiz-Camps I, Del Pozo JL, Oltolini C, DeVoe C, Drgona L, Gasch O, Mikulska M, Martin-Davila P, Peghin M, Vazquez L, Laporte-Amargos J, Dura-Miralles X, Pallares N, Gonzalez-Barca E, Alvarez-Uria A, Puerta-Alcalde P, Aguilar-Company J, Carmona-Torre F, Clerici TD, Doernberg SB, Petrikova L, Capilla S, Magnasco L, Fortun J, Castaldo N, Carratala J, Gudiol C. Real-Life Use of Ceftolozane/Tazobactam for the Treatment of Bloodstream Infection Due to Pseudomonas aeruginosa in Neutropenic Hematologic Patients: a Matched Control Study (ZENITH Study). Microbiol Spectr. 2022 Jun 29;10(3):e0229221. doi: 10.1128/spectrum.02292-21. Epub 2022 Apr 27. PMID 35475683